CLINICAL TRIAL: NCT06235164
Title: The Safety and Efficacy of Neoadjuvant Immunochemotherapy Followed by Laparoscopic Gastrectomy for Gastric Cancer: A Multicenter Real-world Clinical Study
Brief Title: The Safety and Efficacy of Neoadjuvant Immunochemotherapy Followed by Laparoscopic Gastrectomy for Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Fujian Medical University Union Hospital, Fujian Medical University
Other Study IDs: 2023KY160
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Locally Advanced Gastric Cancer
MeSH Terms: interventions — Nivolumab; camrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neoadjuvant immunochemotherapy group: The immune checkpoint inhibitors (ICIs) used for neoadjuvant immunotherapy in this study included sintilimab, nivolumab, and camrelizumab. Neoadjuvant chemotherapy regimens were primarily categorized into two- and three-agent regimens. The two-agent regimens included: SOX (S-1 + oxaliplatin), CapeOx (capecitabine + oxaliplatin), AS (S-1 + nab-paclitaxel), FOLFOX (oxaliplatin + fluorouracil) and DS (S-1 + docetaxel). The three-agent regimens included: FLOT (docetaxel + oxaliplatin + fluorouracil), DOS (docetaxel + oxaliplatin + S-1) and POF (paclitaxel + oxaliplatin + fluorouracil). Dosages were calculated based on drug monographs, guidelines, and patient body surface area. The patients underwent LG within 4-6 weeks after completing neoadjuvant therapy.
  Interventions: Drug: immune checkpoint inhibitors: sintilimab, nivolumab, and camrelizumab
- neoadjuvant chemotherapy group: Neoadjuvant chemotherapy regimens were primarily categorized into two- and three-agent regimens. The two-agent regimens included: SOX (S-1 + oxaliplatin), CapeOx (capecitabine + oxaliplatin), AS (S-1 + nab-paclitaxel), FOLFOX (oxaliplatin + fluorouracil) and DS (S-1 + docetaxel). The three-agent regimens included: FLOT (docetaxel + oxaliplatin + fluorouracil), DOS (docetaxel + oxaliplatin + S-1) and POF (paclitaxel + oxaliplatin + fluorouracil). Dosages were calculated based on drug monographs, guidelines, and patient body surface area. The patients underwent LG within 4-6 weeks after completing neoadjuvant therapy.

INTERVENTIONS:
Drug: immune checkpoint inhibitors: sintilimab, nivolumab, and camrelizumab — Drug: Sintilimab, Nivolumab, and Camrelizumab，One course will last 21 days.Given once every 3 weeks at a dose of 200 mg. Drug: nab-paclitaxel nab-paclitaxel one course will last 21 days#Given twice every 3 weeks at a dose of 125 mg/m2. Drug:oxaliplatin Oxaliplatin one course will last 21 days#Given once every 3 weeks at a dose of 130 mg/m2.
  Drug:docetaxel docetaxel one course will last 21 days#Given once every 3 weeks at a dose of 40mg/m2.
  Drug:fluorouracil fluorouracil one course will last 14 days#Given once every 2 weeks at a dose of 2800mg/m2.
  Drug: Capecitabine Capecitabine was calculated according to body surface area every 3 weeks at a dose of 1000 mg/m2, P.O., bid, d1-d14 Drug: S1 S-1 was calculated according to body surface area, P.O., bid, d1-d14#And the dosage according body surface area:<1.25m2, 40mg everytime;1.25-1.5m2,50mg every time; >1.5m2, 60mg every time
  Groups: neoadjuvant immunochemotherapy group

SUMMARY:
To evaluate the safety and effectiveness of laparoscopic gastrectomy (LG) following neoadjuvant immunochemotherapy (nICT)

DETAILED DESCRIPTION:
comparing the radiological response, pathological response rate, perioperative outcomes, and early recurrence between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-85 years of age
* Gastric adenocarcinoma was confirmed by pathology# including histology or cytology##
* CT/MRI,PET-CT or laparoscopic exploration were used to confirm the diagnosis of gastric cancer staging as cT2-4a and/or N+ and M0 before operation.
* measurable lesions at least should be detected by CT/MRI examination in accordance with the RECIST1.1.#CT scan of tumor lesion length≥10mm#CT scan short diameter≥15mm#scan slice thicknes 5mm#
* ECOG#Eastern Cooperative Oncology Group#PS#Performance Status#:0-1 scores;
* the expected survival time is more than 12 weeks
* the main organ function is normal, which should meet the following criteria:

  (1) blood routine examination standards should be met#no blood transfusion within 14 days#

  a#HB≥ 100g/L b. WBC≥3×109/L c. ANC≥1.5×109/L d. PLT≥100×109/L #2#biochemical examination shall comply with the following criteria#
  1. BIL#1.5 normal upper limit ULN
  2. ALT and AST#2.5 ULN,GPT≤1.5×ULN
  3. Cr≤1 ULN#CCR#creatinine clearance rate#60ml/min(Cockcroft Gault formula)
* women of childbearing age must have a pregnancy test in 7 days before entering the group (in serum), and the results were negative, and willing to use appropriate contraception during the study period and the last 8 weeks after giving drug test; men should have the surgical sterilization, or adopt the appropriate contraceptive methods during the test and the last 8 weeks after giving drug test#
* No other clinical studies were conducted before and during the treatment
* participants is willing to participate in this study, sign the informed consent, have good compliance, cooperate with follow-up.

Exclusion Criteria:

* Previous history of chemotherapy, radiotherapy, targeted drug therapy or immunotherapy
* Patients with contraindications for surgical treatment and chemotherapy or whose physical condition and organ function do not allow for larger abdominal surgery
* patients with metastasis
* Having any active autoimmune diseases or a history of autoimmune diseases (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); Patients with vitiligo or cured childhood asthma/allergies who did not need any intervention in adulthood were excluded; Autoimmune hypothyroidism treated with a stable dose of thyroid replacement hormone; Type 1 diabetes with stable doses of insulin
* A history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency disorders, or a history of organ transplantation and allogeneic bone marrow transplantation
* Accompanied by serious heart, lung, liver, kidney disease; Have nerve, mental disease; Jaundice or obstruction of the digestive tract with severe infection
* pregnant or lactating women
* The blood pressure of patients with hypertension cannot be reduced to the normal range by the antihypertensive drugs (systolic pressure >140 mmHg, diastolic pressure >90 mmHg)
* With # magnitude of coronary heart disease, arrhythmia (including QTc protracted between male > 450 ms, women > 470 ms) and cardiac insufficiency
* Patients have a clear tendency with gastrointestinal bleeding, including the following situation: local active ulcerative lesions, and fecal occult blood (+ +); with melena and hematemesis history in 2 months; and patients with fecal occult blood (+) and unresected gastric primary tumor; patients with the risk of bleeding should take the gastroscopy test, if it is the gastric cancer, and researchers believe that may results in massive digestive tract hemorrhage#coagulation dysfunction (INR(international normalized ratio)>1.5, APTT(activated partial thromboplastin time)>1.5 ULN), with bleeding tendency;
* Subjects have failed to control good cardiovascular clinical symptoms or disease, including but not limited to: such as: (1) the NYHA class II heart failure (2) above unstable angina pectoris (3) occurred within 1 year (4) have clinical significance of myocardial infarction (mi) room sex or ventricular arrhythmias without clinical intervention on or after clinical intervention is still poorly controlled
* History of interstitial lung disease (except radiation pneumonia without hormone therapy), and history of non-infectious pneumonia
* Patients are positive of urine protein (urine protein detection 2+ or above, or 24 hours urine protein quantitative >1.0g);
* A person who has previously been allergic to any component of camrilizumab or to any component of the drug under study
* The researchers consider those who were not suitable for inclusion.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with locally advanced gastric cancer who underwent neoadjuvant therapy
Sampling Method: Non-Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
pathological complete response | 4 months
  pathological complete response (pCR)

SECONDARY OUTCOMES:
major pathological response | 4 months
  major pathological response#MPR

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No